CLINICAL TRIAL: NCT05490511
Title: Drug-gene-nutraceutical Interactions of Cannabidiol and Tacrolimus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Michael Eadon, Associate Professor of Medicine, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12763; 5R01AT011463-02 (NIH)
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-06

CONDITIONS: CBD; Transplant Complication; Kidney Disease, Chronic
Keywords: cannabidiol; tacrolimus; CYP3A5
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Tacrolimus; Cannabidiol

STUDY DESIGN:
Intervention Model Description: Subjects participate in a 3-phase fixed sequence pharmacokinetic study to evaluate the interaction between tacrolimus, cannabidiol, and genotype on tacrolimus AUC and immune system pharmacodynamic outcomes. Subjects with and without CKD will be enrolled in parallel arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- CYP3A5 expressers without chronic kidney disease (Active Comparator)
  Interventions: Drug: Tacrolimus single dose; Drug: Epidiolex single dose; Drug: Epidiolex steady-state and tacrolimus single dose
- CYP3A5 non-expressers without chronic kidney disease (Active Comparator)
  Interventions: Drug: Tacrolimus single dose; Drug: Epidiolex single dose; Drug: Epidiolex steady-state and tacrolimus single dose
- CYP3A5 expressers with chronic kidney disease (Active Comparator)
  Interventions: Drug: Tacrolimus single dose; Drug: Epidiolex single dose; Drug: Epidiolex steady-state and tacrolimus single dose
- CYP3A5 non-expressers with chronic kidney disease (Active Comparator)
  Interventions: Drug: Tacrolimus single dose; Drug: Epidiolex single dose; Drug: Epidiolex steady-state and tacrolimus single dose

INTERVENTIONS:
Drug: Tacrolimus single dose — 5 mg once
  Other Names: Period 1
Drug: Epidiolex single dose — Epidiolex 5 mg/kg
  Other Names: Period 2
Drug: Epidiolex steady-state and tacrolimus single dose — Epidiolex at up to 5 mg/kg twice daily (for 14 days) and tacrolimus 5 mg once on day 12 of period
  Other Names: Period 3

SUMMARY:
The information learned in these studies will help to inform doctors as to how to appropriately adjust doses of cannabidiol and tacrolimus in order to improve health outcomes and long-term treatment success for transplant recipients.

DETAILED DESCRIPTION:
The commercial availability of cannabidiol, or CBD oil, has increased in the United Stated and this supplement has the potential to cause a variety of drug-drug interactions, including in solid organ transplant recipients who receive tacrolimus to prevent rejection. Through a series of pharmacokinetic and pharmacodynamics assays, this proposal will identify gene-drug and drug-drug interactions (DDI), including those that place transplant recipients at risk for increased toxicity related to their immunosuppression. The information learned in these studies will help to inform practitioners as to whether cannabidiol needs to be avoided in transplant recipients and how to appropriately adjust doses of CBD and immunosuppression in order to improve health outcomes and long-term treatment success in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Are judged healthy enough to participate as determined by and decided from a pre-enrollment screening session that includes medical history and laboratory tests such as blood and urine tests, and electrocardiography (EKG).
* Agree to refrain from taking any prescription medications, over-the-counter medications, and herbal, dietary, and alternative supplements that may interact with the metabolism of the study drugs at least 2 weeks prior to the start of the study and until study completion.
* Are willing to commit the time requested for this study
* Are willing to refrain from smoking or use of tobacco or marijuana for at least two weeks prior to and until the completion of the study (the entire study lasts for approximately 26 days).

Additional Criteria for the Healthy volunteer study:

• Have a GFR above 60 ml/min/1.73m2 with proteinuria less than 0.3 grams by urine protein to creatinine ratio or 24 hour urine collection

Additional Criteria for the CKD study:

* Have either:
* A GFR less than or equal to 60 ml/min/1.73m2 or
* The presence of greater than 0.3 grams of proteinuria by urine protein to creatinine ratio or 24 hour urine collection, but less than 3.5 gm of nephrotic range proteinuria as hypoalbuminemia may impact protein binding.

Exclusion Criteria:

* Unable to provide informed consent
* Have history of intolerance, allergic reactions (e.g. rash) or other forms of hypersensitivities to any of the study medications (tacrolimus or cannabidiol);
* Are currently taking sedative agents, including agents for insomnia
* Are underweight (body mass index (BMI) less than 18.5) or overweight [body mass index (BMI) greater than 35]
* Have a positive pregnancy serum or urine test obtained just prior to each study, or are breast feeding
* Are night shift workers
* Are on dialysis
* Have compromised liver function as defined by pre-screening bilirubin, AST and ALT testing including any elevation of bilirubin or AST/ALT more than 2x the upper limit of normal.
* Are not willing to refrain from smoking or use of marijuana for at least two weeks prior to and until the completion of the study
* Have a Hgb < 10.0 g/dL
* Have gastrointestinal (digestive) disorders such as persistent diarrhea or malabsorption that would interfere with the absorption of orally administered drugs
* Have a history of or current seizure disorder
* Are currently on immunosuppression or are immunosuppressed.
* Are recipients of a current allograft (heart, kidney, pancreas, liver, intestine, lung, stem cell transplant).
* Have baseline EKG readings that are abnormal that could place the patient at the high risk.
* Have alcohol (more than 4 alcoholic drinks per day on a regular basis) or drug abuse, including opioids, or have used tobacco products or marijuana within the past three months, and are unwilling or unable to stop taking these medications two weeks prior to and during the entire study period
* Have participated in a research study involving intensive blood sampling or have donated blood within the past two months
* Had an unplanned hospitalization in the last 6 months or two or more unplanned hospitalizations in the last 2 years.
* Are taking prescription medications, that may interfere with the metabolism of the study drugs (e.g., inhibitors or inducers of CYP3A4/5 or CYP2C19 or those that will displace protein binding of tacrolimus/cannabidiol). Interactions will be screened according to the Flockhart table.
* Are taking over-the-counter medications, herbal or dietary supplements, and alternative medicines that may interfere with the metabolism of the study drugs (e.g., inhibitors or inducers of CYP3A4/5 or CYP2C19 or those that will displace protein binding of tacrolimus/cannabidiol) that the subject is unwilling or unable to stop over the course of the study. Interactions will be screened according to the Flockhart table.
* Are students under supervision of any of the study investigators.
* Cannot commit the time requested for this study.
* Have a known CYP3A4 *22/*22 genotype

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2025-08-31 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
The AUC0-Infinity ratio of tacrolimus with cannabidiol divided by tacrolimus alone | 27 days
  The primary outcome is the AUC0-Infinity ratio of tacrolimus with cannabidiol divided by tacrolimus alone between CYP3A5 expressers and non-expressers in subjects with and without chronic kidney disease (CKD). Subjects with and without CKD will be analyzed separately.

SECONDARY OUTCOMES:
Immune cell distribution and signaling as measured by scRNA sequencing | 27 days
  Immune cell distribution and signaling as measured by scRNA sequencing. The hypothesis tested is that cannabidiol will induce T regulatory lymphocytes (Tregs) and reduce overall cytokine signaling as compared to tacrolimus alone. Period 1 and Period 3 will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Eadon, MD, Principal Investigator — Indiana University School of Medicine; Zeruesenay Desta, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- IU Health University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Birdwell KA, Decker B, Barbarino JM, Peterson JF, Stein CM, Sadee W, Wang D, Vinks AA, He Y, Swen JJ, Leeder JS, van Schaik R, Thummel KE, Klein TE, Caudle KE, MacPhee IA. Clinical Pharmacogenetics Implementation Consortium (CPIC) Guidelines for CYP3A5 Genotype and Tacrolimus Dosing. Clin Pharmacol Ther. 2015 Jul;98(1):19-24. doi: 10.1002/cpt.113. Epub 2015 Jun 3. PMID 25801146
- [Background] Brown JD, Winterstein AG. Potential Adverse Drug Events and Drug-Drug Interactions with Medical and Consumer Cannabidiol (CBD) Use. J Clin Med. 2019 Jul 8;8(7):989. doi: 10.3390/jcm8070989. PMID 31288397
- [Derived] Gisch DL, Koyama S, Etkins J, So GC, Fehrenbach DJ, Lu JBL, Cheng YH, Ferreira RM, Rajadhyaksha E, McClara K, Asghari M, Sharfuddin AA, Dagher PC, Snell LM, Madhur MS, Polidoro RB, Desta Z, Eadon MT. Cannabidiol exerts antiinflammatory effects but maintains T effector memory cell differentiation in humans. JCI Insight. 2025 Nov 18;11(1):e198590. doi: 10.1172/jci.insight.198590. eCollection 2026 Jan 9. PMID 41252210